CLINICAL TRIAL: NCT01331603
Title: Assessment of Labile Plasma Iron (LPI) as an Alternative Parameter for Iron Overload in MDS and Primary Myelofibrosis Patients With Iron Overload and Its Correlations With the Classical Iron Overload Parameters.
Brief Title: Assessment of Labile Plasma Iron (LPI) in Myelodysplastic Syndromes (MDS) and Primary Myelofibrosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Dr' Ghoti Hussam, Hematology department of Wolfson Medical Center
Other Study IDs: LPI1CTIL
Record Dates: First submitted 2011-01-18; First posted 2011-04-08 (Estimated); Last update posted 2011-04-08 (Estimated); Status verified 2011-03

CONDITIONS: Myelodysplastic Syndrome; Primary Myelofibrosis
Keywords: MDS; primary myelofibrosis; low+high risk MDS patients; patients
MeSH Terms: conditions — Myelodysplastic Syndromes; Primary Myelofibrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- MDS and primary myelofibrosis patients: patients with in iron overloaded MDS patients (low and high risk ), and also patients with primary myelofibrosis. The risk stratification of these patients will be calculated according to the IPSS (International Prognostic Scoring System).

SUMMARY:
Recently, it has been demonstrated that iron overload is associated with the appearance of labile plasma iron (LPI).

LPI is redox active and is rapidly taken up by cells, leading to a rise in the labile iron pool (LIP) and catalyzing generation of reactive oxygen species (ROS), which can lead to cellular damage.

The LPI data are mostly derived from thalassemia iron overload research , however, there are a few data describing LPI and its correlations with the classical iron overload parameters (ferritin, TSAT) in acute anemias such as MDS Therefore we are going to assess LPI in iron overloaded myelodysplastic syndromes (MDS) (low and high risk) and primary myelofibrosis, in order to assess whether it can be used as alternative to the routinely used parameters; TSAT and ferritin levels.

DETAILED DESCRIPTION:
Approximately 60-80% of patients with myelodysplastic syndromes (MDS) present with symptomatic anemia and 80-90%, of these, will require red blood cell (RBC) transfusions. Excess transfusional iron causes iron overload (IO) which is characterized by elevated serum ferritin (> 1000ng/ml) and transferrin saturation (TSAT > 50%) levels.

Assessment of IO using serum ferritin and TSAT levels is not accurate enough and this is due to changes in serum ferritin and TSAT during any inflammatory condition.

Since serum ferritin is considered as a positive acute phase reactant and therefore inflammatory state can lead to an increase in serum ferritin levels and so does not reflect the exact amount of iron overload.

In contrast TSAT can decrease during inflammation and in addition it follows diurnal variations.The aim of our present study is to asses the levels of LPI in patients with in iron overloaded MDS patients (low and high risk), and also patients with primary myelofibrosis, in order to find out any laboratory correlations between LPI, TSAT and srum ferritin levels.

Methods:

The study will contain 50 patients low+high risk MDS patients and patients with primary myelofibrosis with iron overloaded. The risk stratification of these patients will be calculated according to the WPSS (WHO adapted Prognostic Scoring System)

After ICF (Informed Consent Form) has been signed by the patients the following laboratory tests will be taken once during the study:

* Ferritin (local laboratory)
* Transferrin Saturation (local laboratory)
* CRP (local laboratory)
* LPI (feROS™ eLPI from Aferrix Ltd., Tel- Aviv, Israel)

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years old
* MDS patients (low and high risk )

Exclusion Criteria:

* age < 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: low and high risk MDS patients and primary myelofibrosis patients.The risk stratification of these patients will be calculated according to the WPSS (WHO adapted Prognostic Scoring System)
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2011-03; Primary Completion 2013-01 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
The value of Ferritin,Transferrin Saturation,CRP and LPI at the blood samples | 1 year
  The blood samples should be taken at least one week apart from last blood transfusion.
  In case of infection or acute inflammation , blood samples should be taken only one week after resolution of these conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Ghoti Hussam, MD, Principal Investigator — Hematolgy Department of Wolfson Medical Center
Locations (1):
- Wolfson Medical Center, Holon, Israel